CLINICAL TRIAL: NCT00317655
Title: Glucosamine Sulphate, Ginger, Ginger-Avocado-Soya and Ginger-Ibuprofen for Chronic Back Pain - a Randomized, Double Blind, Placebo-Controlled Clinical Investigation With Parallel Groups for 3 Months to Enlighten Joint Health
Brief Title: Glucosamine Sulphate, Ginger, Ginger-Avocado-Soya and Ginger-Ibuprofen for Chronic Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferrosan AS (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jointcare/Fe/1/DK; Eudractnr. 2005-002691-15
Record Dates: First submitted 2006-04-23; First posted 2006-04-25 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Back Pain
Keywords: back pain
MeSH Terms: conditions — Back Pain | interventions — Glucosamine; ginger extract

INTERVENTIONS:
Drug: Glucosamine sulphate
Drug: Ginger
Drug: Ginger-Avocado-Soya
Drug: Ginger-ibuprofen

SUMMARY:
The main purpose of this study is to investigate the ability of some dietary supplement products to affect general joint health and life quality in a selected population with back pain.

The study is randomized and double - blind, with parallel groups receiving treatment for a duration of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic back pain daily or almost daily for at least 3 months prior to inclusion
* Patient classified as I or II according to Quebec Task Force
* No intake of glucosamine sulphate, ginger, or avocado-soya extract during last 3 months
* Fertile women should, at start, have a negative pregnancy test and during test use acceptable prevention methods (p-pills, intrauterine device [IUD], depot gestagen, subdermal implant, hormonal vaginal ring or transdermal depot plaster).
* Anxiolytics, muscle relaxants, physiotherapy, chiropractic treatment, or training should not have been used during last 3 months.

Exclusion Criteria:

* Serious disease (eg. heart disease, cancer (within past 5 years), kidney disease, blood diseases, inflammatory diseases (eg. chronic rheumatoid arthritis, fibromyalgia)
* Suspicion that back pain is caused by osteoporosis, other arthritic condition than osteoarthritis, cancer, infection, pain from organ disease or psychosomatic cancer disease.
* Uncontrolled elevated blood pressure, defined as systolic ≥ 160 mm Hg or diastolic ≥ 90 mm Hg.
* VAS measurement at inclusion less than ved 30 mm or over 90 mm.
* Prehistory of ulcer, stomach surgery, or inflammatory bowel disease
* Pain relief medication besides must not be taken during study.
* Patients in need of non-steroidal anti-inflammatory drugs (NSAIDs), morphine, or similar medication are not eligible. Same is also valid for patients in need of injections or acupuncture.
* Back surgery within 6 months before inclusion or earlier surgery without effect
* "Heart" aspirin (low dose), ulcer medication, or blood thinning medication
* Alcohol abuse
* Depression
* Pregnancy or breastfeeding
* Allergy to crustaceans or known intolerance for glucosamine sulphate, ginger, avocado, soy, or ibuprofen
* Allergy or asthma released by salicylic acid or other arthritis medication (NSAIDs)
* Patient who is seeking pension due to back pain or has other economical interests connected to his/her back pain

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2006-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
mm pain relief (visual analog scale [VAS]) during past 24 hours compared from start (0 weeks) and 12 weeks

SECONDARY OUTCOMES:
Percentage of responders showing more than 15 mm improvement in pain relief
mm pain relief (VAS) within past 7 days at weeks 1, 2, 4, 6, 9, and 12
Function level according to Roland Morris-questionnaire (23 points)
Patients' Global Impression of Change (pain)
Patients' satisfaction with pain medication
Use of rescue medication
Adverse events profile
Body weight (start and 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Keld Østergaard, MD, PhD, Principal Investigator — Slidgigtinstituttet A/S
Locations (1):
- Slidgigtinstituttet A/S, Ishøj, Denmark